CLINICAL TRIAL: NCT06258850
Title: REstoration With Calcifediol of VItamin D Deficiency in Pulmonary Arterial Hypertension Patients
Brief Title: REstoration of VItamin D in Pulmonary Arterial Hypertension
Acronym: REVIDAH
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Universidad Complutense de Madrid (Other); Hospital Clinic of Barcelona (Other); Hospital Vall d'Hebron (Other); Hospital Universitario Marqués de Valdecilla (Other); Hospital Universitario de Gran Canaria Doctor Negrín (Unknown); Hospital Universitario La Fe (Other); Hospital Universitario Doctor Peset (Other); Hospital Universitario Ramon y Cajal (Other); Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Principal Investigator, Diego Agustín Rodríguez, MD, PhD. Head of Pneumology Department, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICI23/00001
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Pulmonary Artery Hypertension; Vitamin d Deficiency
Keywords: Clinical improvement; Clinical worsening
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension; Vitamin D Deficiency | interventions — Calcifediol; Vitamin D

STUDY DESIGN:
Intervention Model Description: Multicenter clinical trial, placebo-controlled, randomized (1:1 ratio), in two parallel groups (without crossover), cuadruple blind, and add-on on existing treatments.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo capsules will be identical to those of the active treatment. The batch of capsules for each patient will be codified and codes will be provided by the producing company to the SCReN platform who will keep them so that patients and investigators and the local pharmacy will be blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Calcifediol (Experimental): Calcifediol (25-OH vitamin D3) in oral soft capsules (Hidroferol® 0,266 mg, equivalent to 15960 IU vitamin D).
  Interventions: Drug: Calcifediol Oral Capsule
- Placebo (Placebo Comparator): Placebo in oral soft capsules (externally indistinguishable from Hidroferol®).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Calcifediol Oral Capsule — One Hydroferol® soft capsule (0.266 mg) will be administered once weekly for the first 12 weeks and one capsule every two weeks for the next 12 weeks.
  Other Names: Vitamin D
  Arms: Calcifediol
Drug: Placebo — One soft capsule will be administered once weekly for the first 12 weeks and one capsule every two weeks for the next 12 weeks.
  Other Names: Control
  Arms: Placebo

SUMMARY:
Background. Pulmonary arterial hypertension (PAH) is a heterogeneous pathophysiological condition characterized by progressive pulmonary vascular narrowing that ultimately results in right-sided heart failure and eventually death or lung transplantation. The effectiveness of current pharmacological treatments is suboptimal and a large proportion of patients still had events or died despite receiving combination therapy. Vitamin D deficiency has been found to be much more frequent in PAH patients than in the general population or even compared to patients with other severe cardiovascular diseases. Moreover, vitamin D deficiency has a negative prognostic impact in PAH. Animal studies support that vitamin D deficiency worsens PAH.

Hypothesis. In patients with PAH and vitamin D deficiency, restoration of vitamin D status with calcifediol improves their symptomatology and prognosis.

Design: Multicenter clinical trial with the participation of 9 hospitals, placebo-controlled, randomized (1:1 ratio), in two parallel groups (without crossover), triple blind, and add-on on existing treatments (add-on). It will include at least 102 subjects (51 in the calcifediol group and 51 in the placebo group) followed for 24 weeks of treatment.

Inclusion criteria: Patients of both sexes (18-75 years) with hemodynamic diagnosis of PAH and severe vitamin D deficiency (25-OHvitD <= 12 ng/ml) and without previous diagnosis of osteoporosis or osteomalacia.

Treatments: 1) Calcifediol Hydroferol® 0.266 mg once every 10 days for the first 12 weeks and once every two weeks for the following 12 weeks. 2) Placebo.

Main objective: A composite endpoint of clinical improvement without clinical worsening at week 24.

Expected outcome: Restoration of vitamin D status is an unexpensive measure, very easily implantable and that could improve the evolution of the disease as well as other aspects such as bone or immune health and that has few side effects.

DETAILED DESCRIPTION:
RESEARCH TEAM PI: Diego A. Rodríguez Chiaradía, Co-PI: Francisco Perez-Vizcaino. Investigators: Joan A. Barberá, Isabel Blanco Vich, Manuel Lopez Meseguer, Amaya Martinez Menaca, Gregorio M Perez Peñate, Raquel López Reyes, Alberto García Ortega, Jose Andres Tenes, Remedios Otero.

RATIONALE: There is no evidence to support that there is a causal link, at least in humans, between vitamin D deficiency and PAH. Moreover, if present, the causal relationship might be in either direction: vitamin D causing/aggravating PAH or PAH inducing vitamin D deficiency. Only data from preclinical or small uncontrolled trials are available that suggest that low vitamin D aggravates PH. Thus, the key clinical question for PAH patients that we are addressing herein is: Does restoration of vitamin D levels lead to clinical improvement and better prognosis in PAH patients?

Thus, our HYPOTHESIS is that in patients with stable PAH and vitamin D deficiency, restoration of the vitamin D status with calcifediol supplements improves symptoms and prognosis.

MAIN OBJECTIVE. To analyze whether a vitamin D supplement (0,266 mg calcifediol, once every 10 days for the first 12 weeks and once every second week in the following 12 weeks) induces clinical improvement without clinical worsening at week 24 compared with placebo.

DISEASE. The study will be performed in patients with PAH and severe deficit of vitamin D. Patients will be at intermediate risk of 1-year mortality according to 2022 European Respiratory Society /European Society of Cardiology guidelines despite receiving standard treatment for PAH for at least 6 weeks before randomisation.

CLINICAL PHASE. Phase IV clinical trial analyzing the therapeutic effects, as measured by a composite endpoint of morbidity and mortality, of a commercial source of vitamin D (Hidroferol® 0,266 mg) available in Spain.

PARTICIPATING CENTERS. This is a multicentric study that will be conducted in 9 hospital-based pulmonary hypertension centres in Spain.

ETHICS AND PATIENT CONSENT. The institutional review board at each participating centre will approve the protocol, and the study will be carried out in accordance with Good Clinical Practice guidelines and the Declaration of Helsinki. All patients will provide written informed consent.

STUDY DESIGN. Multicentric, randomized, placebo controlled (1:1 proportion), quadruple blind, parallel, add-on, superiority trial.

EXPERIMENTAL DRUG AND ROUTE OF ADMINISTRATION. Patients in the active arm will receive oral calcifediol (25-OH vitamin D3) or placebo.

DOSING: One Hydroferol® soft capsule (0.266 mg) or one placebo capsule will be administered once every 10 days for the first 12 weeks and one capsule every two weeks for the next 12 weeks.

ADD-ON. At randomization patients must be treated with the standard care including the specific drugs for PAH according to ERS/ESC guidelines and stable for at least 6 weeks. Patients will start the active or placebo treatment and remain with their current PAH treatments.

STUDY POPULATION: Patients of both sexes and ages between 18 years and 75 years with a diagnosis of PAH and severe vitamin D deficiency.

PATIENT RECRUITMENT. Patients with a previous diagnosis of PAH, stable for the 6 weeks, that regularly attend the PH patient outclinic of the participating hospitals will be recruited.

DIAGNOSIS of PAH. PAH diagnosis according to the 2022 European Society of Cardiology/European Respiratory Society guidelines must have been performed in an accredited PH reference unit. Therefore, patients must present precapillary PH with hemodynamic parameters, measured by right heart catheterization, of mPAP >20 mmHg, pulmonary artery wedge pressure (PAWP) ≤15 mmHg and pulmonary vascular resistance (PVR) >2 WU)] in the absence of other causes of pre-capillary PH, such as chronic thromboembolic PH and PH associated with lung diseases.

DEFINITION OF SEVERE VITAMIN D DEFICIENCY. The best biomarker of vitamin D status is the serum or plasma level of the hydroxylated form or vitamin D, 25(OH)-cholecalciferol, also known as 25(OH)-vitamin D or calcifediol. Although there is no universal consensus on its optimal levels or those representing insufficiency or deficiency, most scientific societies and regulatory agencies define vitamin D deficiency as serum or plasma levels of 25(OH)-vitamin D below 20 ng/ml. According to this, ninety-five percent of the patients with PAH in the Spanish cohort showed vitamin D deficiency. However, patients with the lowest values showed poorer prognosis, suggesting that there are important differences depending on the severity of the deficit. Therefore, patients with the most severe deficiency are expected to be those obtaining greatest benefit. There is no widely accepted definition of severe deficiency. Herein, we will define severe vitamin D deficiency as serum 25(OH)-vitamin D levels equal to or less than 12 ng/ml. According to this definition and the data of the Spanish PAH cohort, we expect that ~75% of the otherwise eligible PAH patients will fit into this category. This arbitrary cutoff value intends to recruit a large percentage of patients that are expected to have the maximal benefit. Therefore, patients with values of 12-20 ng/ml that would potentially obtain marginal benefit will be excluded.

RANDOMIZATION. Patients will be randomized 1:1 to placebo (the control arm) or to Hidroferol (active arm). A randomization list will be generated using the SAS 9 software for Windows. The randomization list will be imported into the REDCap program so that researchers can randomize candidate subjects using a more user-friendly interface. Subjects who meet the selection criteria will be randomized between treatment groups, in order to achieve balanced randomization in treatment groups. The treatment assignment will be centralized, thus keeping the sequence hidden.

BLINDING AND MASKING. Placebo capsules will be identical to those of the active treatment. The batch of capsules for each patient will be codified and codes will be provided by the producing company to the SCReN platform who will keep them so that patients and investigators, the local pharmacy will be blind.

MAIN VARIABLES OF THE STUDY. Baseline and 6-month values of the following variables will be compared and be used either for the composite endpoint or as secondary objectives: a) 6MWD, b) serum pro-BNP, c) functional class (WHO/NYAS), d) noninvasive risk score (NIRS) based on the three previous variables, e) ventricular function analyzed echocardiographically by TAPSE and f) a mechanistic parameter: serum noggin levels (difference: at 6 months minus baseline). In addition, quality of life will be compared using the emPHasis-10 questionnaire. Echo-doppler will be performed at each hospital and the images will be centrally and blindly analyzed by a single expert echocardiographer.

VISITS. Visit 0 (-2 to -4 weeks): Informed consent and eligibility criteria, 6MWD, functional class and blood sampling for 25(OH) vitamin D and NT-proBNP. Visit 1 (week 0): Randomization. Visit 2 (week 12): Safety analysis of 25(OH)vitamin D and calcium levels. Visit 3 (week 24): analysis of efficacy. Central phone calls at week 2, 4, 10 and 20 will be made to assess compliance and possible adverse effects.

WITHDRAWAL OF PATIENTS FROM THE STUDY. Patients must be withdrawn from study treatment: 1) at their own request, 2) when in the investigator's opinion, continuation of the study treatment would be harmful to the patient's well-being. 3) Occurrence of adverse events (AEs) or intercurrent diseases which the investigator judges unacceptable for continuation of participation in the study. 4) Occurrence of adverse drug reactions, which have from the investigator's point of view, a negative impact on the patient's individual risk-benefit ratio. 5) Pertinent noncompliance with the conditions for the study or instructions by the investigator 6) In case of pregnancy or breast feeding 7) Participation in another clinical study, 8) Patient does not tolerate the experimental drug. 9) Patients in the active arm with 25 (OH) vitamin D levels below 20 ng/ml or above 100 ng/ml and patients in the placebo arm with values above 20 ng/ml in the intermediate safety analysis.

RISKS. Adverse reactions of hydroferol® are generally uncommon (> 1/1,000 to < 1/100) although they are sometimes moderately important. The most significant adverse effects are related to excessive intake of vitamin D, especially when associated with high doses of calcium, which is not the case per study protocol. The most characteristic adverse reactions are due to the hypercalcaemia.

INTERMEDIATE SAFETY ANALYSIS. Serum 25(OH)vitamin D will be centrally analyzed in patients receiving either the active treatment or placebo at 12 weeks. The results will be communicated neither to patients nor investigators except for the following cases. Patients in the active arm with 25(OH) vitamin D levels below 20 ng/ml or above 100 ng/ml or with hypercalcemia and patients in the placebo arm with values above 20 ng/ml will be discontinued from the study.

STATISTICAL ANALYSIS Sample size. Calculations for the present project are based mainly in the REPLACE trial (PMID: 33773120). The main endpoint in both trials is similar except that clinical improvement is based on two out of four variables (now includes TAPSE/PASP) instead of two out of three. We expect that this would lead to an increase in events of 25% in both arms. We assume that our placebo group is similar to the REPLACE control group and we expect that the vitamin D group would lead to a clinical improvement similar to that of the riociguat group in REPLACE. The rate of clinical improvement without clinical worsening at week 24 was estimated to be 50% for the vitamin D group and 25% for the placebo. A sample size of 51 patients per arm was calculated using granmo® software (with two-sample frequency, X² test, one-sided alpha=0.05, power=0.8) with an estimated dropout rate of 10%.

Outcomes. All analyses will be performed using the program applied to the SAS statistics, version 9 of the SAS system for Windows. At the end of the study, summaries of the demographic variables and other characteristics of the subjects specified in the data collection notebook will be made according to the two treatment groups. Unless otherwise specified, all continuous variables shall be summarized using number of patients (n), mean, standard deviation, median, minimum, and maximum. Categorical variables shall be described by absolute and relative frequency. The statistical analysis plan (SAP) will be developed and finalized prior to the publication of the database and will describe the populations of subjects to be included in the analyses and the procedures for accounting for missing, unused and non-essential data. Comparisons between groups will be made using one-sided Fisher's exact test. Likewise, a multivariate analysis of the main outcome will be made using a binary logistic regression analysis. Changes on detailed parameters on secondary objectives, will be analyzed through suitable methods for repeated measures (paired t test or equivalent non-parametric Wilcoxon Rank-Sum test). Also, between group differences, will be performed comparing 24 week vs. baseline differences by group. This will be checked through t test or Mann-Whitney test depending on the results of the normality tests in the continuous variables. Finally, repeated measures ANCOVA will be applied to check effects of possible confounding variables.

Data Management Plan. All the data of the participants related to the study will be recorded in an Electronic Data Collection (EDC) whose preparation and maintenance will be carried out from the ISCIII Support Platform for Clinical Research (SCReN).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18 -75 years.
2. Patients with diagnosis of PAH of the following types according to 2022 ERS/ESC guidelines: idiopathic, hereditary, drug and toxin-induced PAH or associated to connective tissues disease.
3. Patients who are stable and treated with standard medications for PAH on monotherapy or with combinations of drugs, including calcium channel blockers, phosphodiesterase type 5 inhibitors (PDE5i), endothelin receptor antagonists (ERA), prostacyclin analogues or selexipag or with stable dose of diuretics who had no treatment modification for at least 6 weeks before randomization.
4. Patients with an intermediate-low and intermediate-high risk score according to 2022 ERS/ESC guidelines.
5. Patients with severe deficiency of vitamin D, defined herein as plasma or serum 25(OH)vitamin D levels equal to or lower than 12 ng/ml
6. Patients who can understand and follow instructions, and who are able to participate in the study for the entire study.
7. Patients must have given their written informed consent to participate in the study after having received adequate previous information and before any study-specific procedures.

Exclusion Criteria:

1. Participation in another interventional clinical study within 30 days before screening.
2. Previous randomisation to treatment during this study (no re-randomisation).
3. Pregnant women or breastfeeding women, or women with childbearing potential not using a effective contraception method throughout the study.
4. Patients with a medical disorder, condition, or history of such that would impair the patient's ability to participate in or complete this study, in the opinion of the investigator.
5. Patients with substance abuse (eg, alcohol or drug abuse) within the previous 3 months before and at randomisation.
6. Patients with underlying medical disorders with an anticipated life expectancy <2 years.
7. Patients with a history of severe allergies or multiple drug allergies or with hypersensitivity to the investigational drug or any of the excipients.
8. Patients unable to perform a valid 6MWD test (eg, orthopaedic disease or peripheral artery occlusive disease that affects the patient's ability to walk).
9. Excluded medication/treatment: active treatment with digoxin.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement without clinical worsening | 24 weeks
  Clinical improvement is defined as a change in at least two of the following variables: 1) increase in 6 minutes walking distance (6MWD) >= 10% or more than 30 m, 2) change from intermediate-low or intermediate-high risk to low risk score or change from intermediate-high to intermediate-low risk according to 2022 ERS/ESC guidelines), 3) reduction in BNP or NT-proBNP >= 30%, 4) increase in the TAPSE/SPAP ratio >= 25%. Clinical worsening is defined as any of the following events: a) hospitalization related to PAH, b) therapeutic escalation, c) progression of symptoms, d) lung or cardiopulmonary transplantation, e) atrial septostomy and f) mortality related to PAH.

SECONDARY OUTCOMES:
6 minute walking distance | 24 weeks
  Difference from baseline (active vs placebo)
serum BNP or nt-pro-BNP | 24 weeks
  Difference from baseline (active vs placebo)
functional class (WHO/NYAS) | 24 weeks
  Difference from baseline (active vs placebo)
noninvasive risk score (NIRS) based on the three previous variables | 24 weeks
  Difference from baseline (active vs placebo)
ventricular function analyzed echocardiographically by TAPSE | 24 weeks
  Difference from baseline (active vs placebo)
Serum noggin levels | 24 weeks
  Difference from baseline (active vs placebo)
Quality of life will be compared using the emPHasis-10 questionnaire. | 24 weeks
  Difference from baseline (active vs placebo)

CONTACTS AND LOCATIONS:
Overall Officials: Diego A Rodríguez Chiaradía, MD PhD, Principal Investigator — Hospital del Mar

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with other researcher upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Up to 5 years after the end of the study
Access Criteria: Data will be shared upon request either for collaborative purposes or whenever the researcher has reasonable questions about the study.